CLINICAL TRIAL: NCT02337920
Title: Prediction of Femoral Revascularization Quality Using the Somatic NIRS Signal
Acronym: TEA-NIRS
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: TEA-NIRS
Record Dates: First submitted 2014-11-27; First posted 2015-01-14 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2015-07

CONDITIONS: Lower Limb Vascular Surgery - Femoral Artery Endarteriectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite effective femoral artery endarteriectomy, patients with occlusive arteritis may need complementary stenting of revascularization procedures within the 2 years after the primary surgery because of a poor blood supply in their lower limb extremity. The Near infrared spectrophotometry (NIRS) is a non-invasive monitoring of the brain or tissue oxygenation and provide information on the quality of the local oxygen supply. The aim of our observational study is to correlate the intraoperative NIRS variations at the calf and the soles and the one-year evolution of the arteritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral femoral endarteriectomy

Exclusion Criteria:

* emergency surgery, allergy to adhesive glues, skin abnormalities of the operated leg, multiple associated revascularization procedures other than endarteriectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing unilateral femoral endarteriectomy
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Relationship between the Maximum NIRS difference before and during the femoral artery clamping and the increase of walking perimeter | Change - One month, six months and one year after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Georges Daccache, M.D, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, Calvados, France